CLINICAL TRIAL: NCT04704284
Title: Comparative Analysis of Zero Echo-time MRI and CT for Pediatric Craniosynostosis
Brief Title: Comparing MRI to CT on Pediatric Craniosynostosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Julie B. Guerin, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-007373
Record Dates: First submitted 2020-12-08; First posted 2021-01-11 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Craniosynostosis
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ZTE MRI Imaging (Experimental): Pediatric patients that have gotten a clinically indicated CT within a 6 week time period will receive a Zero Echo Time Magnetic Resonance Imaging (ZTE MRI)
  Interventions: Diagnostic Test: Zero Echo Time Magnetic Resonance Imaging (ZTE MRI)

INTERVENTIONS:
Diagnostic Test: Zero Echo Time Magnetic Resonance Imaging (ZTE MRI) — Magnetic Resonance Imaging (MRI) with zero echo-time (ZTE) that uses proton density differences rather than T2 relaxation time differences to achieve contrast.

SUMMARY:
The purpose of this study is to develop and test the effectiveness and diagnostic quality of Zero Echo Time Magnetic Resonance Imaging (ZTE MRI) in comparison to CT.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 0-18 of age will be recruited by our surgical colleagues based on the clinical concern for craniosynostosis and possible need for calvarial reconstruction.

Exclusion Criteria:

* Lack of consent
* Contraindication/inability to undergo both examinations within the designated time period and/or undiagnostic image quality.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie B Guerin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ZTE MRI Imaging: Pediatric patients that had a clinically indicated CT within a 6 week time period received a Zero Echo Time Magnetic Resonance Imaging (ZTE MRI)
  Zero Echo Time Magnetic Resonance Imaging (ZTE MRI): Magnetic Resonance Imaging (MRI) with zero echo-time (ZTE) that uses proton density differences rather than T2 relaxation time differences to achieve contrast.
Period: Overall Study
Arm/Group | ZTE MRI Imaging
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ZTE MRI Imaging
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.6 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 90% or Greater Concordance Between ZTE and CT Imaging Diagnosis
Description: In the context of our study, concordance refers to the level of agreement between two radiologists in their interpretation of imaging findings across the two modalities (ZTE and CT).
Time Frame: 1 Day
Population: 2 participants data was unanalyzable due to motion artifact.
Measure: Count of Participants; unit: Participants
Arm/Group | ZTE MRI Imaging
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time the participant signed the informed consent form through the end of study completion, approximately 1 day.
Arm/Group | ZTE MRI Imaging
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT04704284/Prot_SAP_000.pdf